CLINICAL TRIAL: NCT02856451
Title: Case Series Analyses of the Risk Factors and Outcomes of Immune-Mediated Encephalitis Following Exposure to Nivolumab
Brief Title: Risk Factors and Outcomes of Immune-Mediated Encephalitis Following Exposure to Nivolumab
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-567
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Encephalitis
MeSH Terms: conditions — Encephalitis | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients Treated with Nivolumab followed by Encephalitis Event: Case series reported to the sponsor from various health care facilities
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days

SUMMARY:
A case series analysis of encephalitis events reported to the Sponsor for patients treated with nivolumab to assess the risk factors and outcomes of immune-mediated encephalitis.

ELIGIBILITY:
Inclusion Criteria:

* Moderate, severe, life-threatening or fatal encephalitis events occurring in patients treated with nivolumab and reported to the Sponsor

Exclusion Criteria:

* Encephalitis cases identified through literature reviews and not reported to the Sponsor
* Encephalitis cases identified from company-sponsored observational studies with secondary data collection
* Spontaneous reports not submitted directly to the Sponsor

Other protocol-defined inclusion/exclusion criteria apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Case series reported to the sponsor from various health care facilities
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Outcomes of Encephalitis | 1 year
  Time since onset of immune-mediated encephalitis to the date of outcome assessment (days) and outcomes defined as: resolved, resolving, death, physical disability (specified), cognitive disability (specified)
Risk factors of Encephalitis | 1 year
  Potential risk factors include but are not limited to medical history including event associated signs/symptoms, and data from brain imaging diffusion, results from lumbar puncture analyses, results from serum sample analyses and results from neurologic examinations

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome